CLINICAL TRIAL: NCT07329725
Title: Impact of Genetic Drivers, Acquired Risk Factors, and Management Strategies on Survival and Clinical Outcomes in Visceral Venous Thrombosis
Brief Title: Genetic Drivers,Risk Factors and Management Strategies on Survival and Clinical Outcomes in Visceral Venous "Thrombosis"
Acronym: Thrombosis
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma mohamed Ahmed Anwer, Principal Investigator, Sohag University
Other Study IDs: Visceral Venous Thrombosis
Record Dates: First submitted 2025-12-23; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Visceral Venous Thrombosis
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort Analysis: Review of medical records to analyze demographic, clinical, and molecular data. Assessment of treatment regimens and outcomes, including thrombotic events, disease progression, and survival rates.
  Interventions: Other: Doppler ultrasonography
- Prospective Cohort Analysis: Consecutive patients will be diagnosed with VVT from [date of ethical approval] forward, enrolled at diagnosis and followed prospectively with standardized baseline testing (including comprehensive genetic panel) and predefined follow-up visits.
  Interventions: Other: Doppler ultrasonography

INTERVENTIONS:
Other: Doppler ultrasonography — Radiological intervention Basic laboratory investigations, and Thrombophilia diagnosis
  Other Names: Chest-X ray; Electrocardiogram (ECG); Echocardiography if indicated.; CT angiography; MR venography; Doppler of the limbs; Basic laboratory investigations; Thrombophilia diagnosis

SUMMARY:
This study aims to evaluate the impact of genetic drivers (somatic and inherited thrombophilias), acquired risk factors, and management strategies on survival and clinical outcomes in patients with VVT using a hybrid prospective-retrospective cohort design.

DETAILED DESCRIPTION:
Observational study (hybrid study comprising a retrospective and prospective cohort analysis):

To evaluate the impact of genetic drivers (somatic and inherited thrombophilias), acquired risk factors, and management strategies on survival and clinical outcomes in patients with VVT using a hybrid prospective-retrospective cohort design.

Data will be collected from the Department of Internal Medicine/hematology unit at Sohag University hospital and clinical databases.

The retrospective component will include eligible patients diagnosed within the preceding ten years, whereas the prospective component will enroll newly diagnosed patients and follow them for one year.

1. Retrospective Cohort Analysis:

   Review of medical records to analyze demographic, clinical, and molecular data. Assessment of treatment regimens and outcomes, including thrombotic events, disease progression, and survival rates.
2. Prospective Cohort Analysis:

Consecutive patients will be diagnosed with VVT from [date of ethical approval] forward, enrolled at diagnosis and followed prospectively with standardized baseline testing (including comprehensive genetic panel) and predefined follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with radiologically confirmed visceral venous thrombosis.
* Availability of complete clinical, laboratory, and imaging data at diagnosis.
* Patients who consent to participate and provide blood samples for genetic testing.

Exclusion Criteria:

* Isolated lower-limb deep-vein thrombosis or pulmonary embolism without visceral involvement.
* Patients with incomplete records precluding outcome assessment.
* Refusal or inability to provide informed consent
* Patients lost to follow-up within the first three months of diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with visceral venous thrombosis, including portal, mesenteric, splenic, renal and hepatic vein thrombosis in Department of Internal Medicine, Sohag University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2025-12-14 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Patients diagnosed with visceral venous thrombosis | The retrospective component will include eligible patients diagnosed within the preceding ten years, whereas the prospective component will enroll newly diagnosed patients and follow them for one year.
  To evaluate the impact of genetic drivers (somatic and inherited thrombophilias), acquired risk factors, and management strategies on survival and clinical outcomes in patients with VVT using a hybrid prospective-retrospective cohort design.

SECONDARY OUTCOMES:
Frequency and distribution | The retrospective component will include eligible patients diagnosed within the preceding ten years, whereas the prospective component will enroll newly diagnosed patients and follow them for one year.
  To estimate the frequency of somatic mutations and inherited thrombophilias and describe their distribution across anatomical sites of VVT (portal, mesenteric, renal, splenic, hepatic) and underlying etiologies (autoimmune, inflammation, cirrhosis, malignancy, post-surgery, idiopathic).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud I Yousef, Associate Prof., Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Boccatonda A, Gentilini S, Zanata E, Simion C, Serra C, Simioni P, Piscaglia F, Campello E, Ageno W. Portal Vein Thrombosis: State-of-the-Art Review. J Clin Med. 2024 Mar 6;13(5):1517. doi: 10.3390/jcm13051517. PMID 38592411
- [Background] Cohen O, Caiano LM, Tufano A, Ageno W. Cancer-Associated Splanchnic Vein Thrombosis. Semin Thromb Hemost. 2021 Nov;47(8):931-941. doi: 10.1055/s-0040-1722607. Epub 2021 Jun 11. PMID 34116580